CLINICAL TRIAL: NCT04608851
Title: Preventing Urinary Tract Infections in Infants and Young Children With Probiotic E. Coli Nissle:
Brief Title: Preventing Urinary Tract Infections With E. Coli Nissle:
Acronym: FinNissle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Turku University Hospital (Other Government); Kuopio University Hospital (Other); Tampere University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Terhi Tapiainen, Adjunct Professor of Pediatrics, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OYS_Tapiainen_002
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Urinary Tract Infections in Children; Secondary Prevention
Keywords: Urinary Tract Infections; E. coli
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: Double Blinded, Placebo controlled and randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention drug or placebo will be given to participants in closed boxes without any labels. Appearance and dosing of the products will be similar. Investigators will not handle the boxes or study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nissle group (Experimental): Intervention will start on the day following the ending of the antimicrobial treatment of the UTI. Patients will receive 1 ml of oral suspension containing 10 E8 CFU/ml of E coli Nissle. Patients under one year of age will receive one daily dose and patients aged more than one year will receive a dose twice daily. Intervention will last for 30 days
  Interventions: Drug: E. coli Nissle
- Control group (Placebo Comparator): Intervention will start on the day following the ending of the antimicrobial treatment of the UTI. Patients will receive 1 ml of oral syrup consisting of Saccharum 630 mg/g and Aqua purificata 370 mg/g. Patients under one year of age will receive one daily dose and patients aged more than one year will receive a dose twice daily. Intervention will last for 30 days
  Interventions: Other: Placebo control

INTERVENTIONS:
Drug: E. coli Nissle — 1 ml of oral suspension containing 10 E8 CFU /ml of E. coli Nissle strain
  Other Names: Mutaflor
  Arms: Nissle group
Other: Placebo control — 1 ml oral syrup consisting of Saccharum 630 mg/g and Aqua purificata 370 mg/g.
  Arms: Control group

SUMMARY:
Urinary tract infections (UTIs) account for 5-14% of pediatric emergency department visits annually. At the moment, up to one third of children suffering of acute (UTI) will have a new infection and there is a lack of effective methods for preventing secondary UTIs in young children. Majority of UTIs in children are caused by intestinal bacteria of the patient, mainly E. coli that colonizes gut of the patient. E. coli Nissle is a probiotic strain that has been used successfully for treating acute gastrointestinal infections in children. The strain has also been proved to be safe for infants and young children. E. coli Nissle could be a potential solution for preventing recurrent urinary tract infections in children as it competes with pathogenic bacteria that usually cause UTIs in children.

The aim of this study is to evaluate efficacy of E. coli Nissle strain in secondary prevention of urinary tract infections in young children.

DETAILED DESCRIPTION:
In order to asses efficacy of E. coli Nissle strain in prevention of recurrent UTIs in children, we aim to conduct randomized, placebo controlled and double blinded clinical trial. We are going to recruit children who are suffering the first urinary tract infection of their life. The UTI will be treated by normal clinical recommendations decided by treating physician. Intervention will start on the day following the last day of the antimicrobial course.

The intervention will last for 15 days and the study participants will receive either intervention drug or placebo. Intervention drug contains 10 E8 CFU/ml of E. coli Nissle strain and will be administered as dose of 1 ml of oral suspension once daily for children aged under one year and twice daily for children aged more than one year.

The study patients will be monitored by monthly electronic surveys for six months after the intervention in order to measure proportion of the children who will have a new UTI during the follow up. We are also going to record possible adverse effects in both study groups. Also use of antimicrobial medication due to any reason will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Children who suffer of the first urinary tract infection of their life defined as pyuria, presence of symptoms (fever or focal symptom), no other explanation for infection, bacterial culture positive or culture result pending
* Written informed consent

Exclusion Criteria:

* Preterm birth, gestational age less than 35 weeks
* Signs of life-threatening infection (such as meningitis)
* Detected anomaly in urinary tract
* Primary immunodeficiency
* Detected anomaly of GE tract
* Ongoing antimicrobial prophylaxis
* Hospital-acquired infection

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 530 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of urinary tract infections | Six months from study entry
  Proportion of the study patient who will have at least one bacterial culture confirmed urinary tract infection

SECONDARY OUTCOMES:
Number of urinary tract infections | Six months from study entry
  Number of bacterial culture confirmed urinary tract infections per person years at risk (PYR)
Hospitalization day due to bacterial culture confirmed urinary tract infection | Six months from study entry
  Number of days spent in the hospital during follow up
Antimicrobial treatment days for suspected or confirmed urinary tract infection | Six months, starting after the initial treatment at study entry has ended
  Number of days when study patient has received antimicrobial treatment
Stomach pain | Six months from study entry
  Number of days with stomach pain reported by families during follow up at web-based surveys
Diarrhea | Six months from study entry
  Number of days with diarrhea reported by families during follow up at web-based survey
Antimicrobial treatment days for any indication | Six months, starting after the initial treatment at study entry has ended
  Number of days when study patient has received antimicrobial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Terhi Tapiainen, MD, PhD, Principal Investigator — University of Oulu
Locations (5):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Department of Pediatrics, Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No
IPD will be shared after reasonable request